CLINICAL TRIAL: NCT03475524
Title: THE METFORMIN AND TRICHLOROACETIC ACID IN TREATMENT OF MELASMA
Brief Title: USE THE SYSTEMIC METFORMIN IN MELASMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karima Nageh, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTM
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study Metformin 1000 mg (Experimental)
  Interventions: Drug: MetFORMIN 1000 Mg Oral Tablet; Drug: Trichloroacetic Acid Peeling
- study Metformin 500 mg (Experimental)
  Interventions: Drug: Trichloroacetic Acid Peeling; Drug: MetFORMIN 500 Mg Oral Tablet
- control group (Placebo Comparator)
  Interventions: Drug: Placebos; Drug: Trichloroacetic Acid Peeling

INTERVENTIONS:
Drug: MetFORMIN 1000 Mg Oral Tablet — oral tablet 1ooomg systemic metformin will be given to group
  Other Names: Glucophage
  Arms: study Metformin 1000 mg
Drug: Placebos — oral placebos will be given to control beside trichloracetic acid peeling
  Arms: control group
Drug: Trichloroacetic Acid Peeling — Trichloroacetic acid peeling to the three groups
Drug: MetFORMIN 500 Mg Oral Tablet — oral tablet 500 mg
  Other Names: Glucophage
  Arms: study Metformin 500 mg

SUMMARY:
Melasma is a chronic and relapsing acquired dyschromia due to an increased epidermal-melanin unit activity that affects sun-exposed areas mainly in women throughout the reproductive years. It is more common in women, accounting for 90% of all cases.The majority of patients are in third and fourth decades of their life. There are several risk factors that influence its appearance including genetic predisposition,exposure to heat and UV radiation, pregnancy, and exogenous hormones (such as oral contraceptives,thyroid hormones, and hormone replacement therapy). Other factors implicated are phototoxic drugs, anticonvulsant medications,and the use of certain cosmetics. Types of melasma are epidermal, dermal and mixed according to location of melanin.

DETAILED DESCRIPTION:
Its pathogenesis is not fully understood, nevertheless there is evidence that melanogenesis in melasma differ from tanning and post-inflammatory hyperpigmentations as well as there is an involvement of the whole epidermal melanin unit in the process (not just hypertrophic melanocytes), mastocytes, fibroblast and endothelium derived cytokines, as well as there are upper dermal abnormalities different from other acquired pigmentary disorders. Patients with melasma have also been found to have higher markers of oxidative stress status.

Melasma has significant impact on patients physical health, interpersonal relationships ,social-well being and self- esteem as they refused to leave their house, felt inferior to others, and incessantly thought about their melasma being.

Melasma is often resistant to treatment and frustrating for both patients and clinician. In spite of presence of several methods for treatment of melasma exacted as, Topical compounds that include the Kligman's formula which is the triple combination of ( retinoid, hydroquinone, and steroid) and azelaic. Chemical peels (e.g., glycolic, β hydroxyl, and trichloroacetic acid )although these must be used cautiously in patients with darker skin. Laser and Light therapies represent potentially promising options for patients who are refractory to other modalities, but they also carry significant risk of worsening the disease.

Recently, some reports refer to the use of metformin in treatment of melasma. Metformin is antidiabetic drugs that was shown to exert its biological effect by decreasing cyclic adenosine phosphate , which is a well known modulator of melanin synthesis. Metformin decreased skin pigmentation in vivo with minimal side effects, suggesting a potential application of metformin in the treatment of hyperpigmentation disorders. Where the metformin was applied topically onto a mouse tail, whitening of the tail was observed. In addition, metformin decreased the epidermal level of melanin when metformin was applied to human skin punch biopsies and to reconstructed human epidermis. When melanocytes were treated with metformin, basal level of total melanin (eumelanin and pheomelanin) were reduced significantly. Also metformin blocked forskolin and alpha melanocyte-stimulating hormone which increase the levels of melanin. Metformin decrease levels of tyrosinase, tyrosinase-related protein-1 and tyrosinase-related protein-2.

ELIGIBILITY:
Inclusion Criteria:

1. All patients above 18 years old with melasma.
2. With Fitzpatrick skin phototypes ranging from Type III-V will recruited.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Current use of hormonal birth control medication or any hormonal therapy, Use of topical hydroquinone within 3 months of study, Use of topical steroids within 1 month of study, Regular use of tanning parlors and History of laser or dermabrasion to the face within 9 months of study.
3. Occupation involving primarily outdoor activities.
4. History of kidney dysfunction diabetic (excluded by history and laboratory), Significant cardiovascular or respiratory disease and any other systemic diseases(i.e,history of endocrine disorders).
5. patients with poor wound healing, recurrent herpes labialis and current skin infection (facial warts, molluscum contagiosum, history of hypertrophic scar/keloids, active dermatosis of atopic, seborrheic or other eczematous type).
6. Photosensitivity,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
degree of improvement of melasma | up to 3 months
  Melasma Area and Severity Index score will be calculated for patients before and after treatment to all patientsscore is calculated by multiplying the area of involvement with the square of pigmentation as given in the formula:
  MSI = 0.4 (a × p 2 ) l + 0.4 (a × p 2 ) r + 0.2 (a × p 2 ) n
  In the formula, "a" stands for "area of involvement," "p" for "severity of pigmentation," "l" for left face, "r" for right face, and "n" for nose.
  The area involved, as well as the severity of pigmentation is scored from 0 to 4Score 0:No visible pigmentation,score 1 :rarely visible pigmentation scor e 2:mild pigmentation score3: moderate pigmentation score 4:sever pigmentation.scoringfor area of involvement less than or equal 10% area involved-scor1,11-30%-score2 ,31-60%-score3 and more than 60%-score 4
  . patient will be photographed at baseline and after every two weeks interval and one month after the last session

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Egypt

REFERENCES:
- [Result] Handel AC, Miot LD, Miot HA. Melasma: a clinical and epidemiological review. An Bras Dermatol. 2014 Sep-Oct;89(5):771-82. doi: 10.1590/abd1806-4841.20143063. PMID 25184917
- [Result] Moubasher AE, Youssef EM, Abou-Taleb DA. Q-switched Nd: YAG laser versus trichloroacetic acid peeling in the treatment of melasma among Egyptian patients. Dermatol Surg. 2014 Aug;40(8):874-82. doi: 10.1097/DSS.0000000000000065. PMID 25068546
- [Result] Brianezi G, Handel AC, Schmitt JV, Miot LD, Miot HA. Changes in nuclear morphology and chromatin texture of basal keratinocytes in melasma. J Eur Acad Dermatol Venereol. 2015 Apr;29(4):809-12. doi: 10.1111/jdv.12453. Epub 2014 Mar 14. PMID 24629163
- [Result] Kong SH, Suh HS, Choi YS. Treatment of Melasma with Pulsed-Dye Laser and 1,064-nm Q-Switched Nd:YAG Laser: A Split-Face Study. Ann Dermatol. 2018 Feb;30(1):1-7. doi: 10.5021/ad.2018.30.1.1. Epub 2017 Dec 26. PMID 29386825
- [Result] Lehraiki A, Abbe P, Cerezo M, Rouaud F, Regazzetti C, Chignon-Sicard B, Passeron T, Bertolotto C, Ballotti R, Rocchi S. Inhibition of melanogenesis by the antidiabetic metformin. J Invest Dermatol. 2014 Oct;134(10):2589-2597. doi: 10.1038/jid.2014.202. Epub 2014 Apr 22. PMID 24756109
- [Result] Sarkar R, Arora P, Garg VK, Sonthalia S, Gokhale N. Melasma update. Indian Dermatol Online J. 2014 Oct;5(4):426-35. doi: 10.4103/2229-5178.142484. PMID 25396123
- [Result] Sheth VM, Pandya AG. Melasma: a comprehensive update: part I. J Am Acad Dermatol. 2011 Oct;65(4):689-697. doi: 10.1016/j.jaad.2010.12.046. PMID 21920241
- [Result] Sheth VM, Pandya AG. Melasma: a comprehensive update: part II. J Am Acad Dermatol. 2011 Oct;65(4):699-714. doi: 10.1016/j.jaad.2011.06.001. PMID 21920242
- [Result] Majid I, Haq I, Imran S, Keen A, Aziz K, Arif T. Proposing Melasma Severity Index: A New, More Practical, Office-based Scoring System for Assessing the Severity of Melasma. Indian J Dermatol. 2016 Jan-Feb;61(1):39-44. doi: 10.4103/0019-5154.174024. PMID 26955093
- [Derived] Ismail SA, Mohamed GA, Mohamedeen KN, Sotohy RSA, Bakr RM. Does Systemic Metformin Have a Role in Treating Melasma? Dermatol Surg. 2024 Apr 1;50(4):366-371. doi: 10.1097/DSS.0000000000004092. Epub 2024 Feb 28. PMID 38416809